CLINICAL TRIAL: NCT01141322
Title: Cholestatic Drug-induced Liver Injury: Correlation With Genotypes of UGT1A1 and 1A7, and Treatment Effect of Ursodeoxycholic Acid
Brief Title: Cholestatic Drug-induced Liver Injury
Acronym: DILI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Yi-Shin Huang, MD, Division of Gastroenterology, Department of Medicine, Taipei Veterans General Hospital, Taipei, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 96-01-23A
Record Dates: First submitted 2010-01-12; First posted 2010-06-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Hepatitis, Toxic
Keywords: drug-induced liver injury; hepatitis, toxic; ursodeoxycholic acid
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UDCA treatment (Experimental): Patients with drug-induced liver injury will be randomly allocated to UDCA treatment group: oral intake ursodeoxycholic acid (UDCA) 13-15 mg/kg BW/day into 3 divided doses after meal till the endpoint or the 8th week. UDCA is 100 mg per tab.
  Interventions: Drug: Ursodeoxycholic Acid
- Placebo (Placebo Comparator): Patients with drug-induced liver injury will be randomly allocated to placebo group. The placebo is of the same color, size and shape as UDCA, and assumed 100 mg per tab. Patients in this group will orally intake 13-15 mg/Kg BW/day of placebo into 3 divided doses after meal as UDCA treatment group, till the endpoint or the 8th week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — ursodeoxycholic acid 13-15 mg/kg BW/day into 3 divided doses after meal till endpoint or the 8th week.
  Other Names: ursodil; UDCA; urso
  Arms: UDCA treatment
Drug: Placebo — The placebo is of the same color, size and shape as UDCA, and assumed 100 mg per tab. Patients in this group will orally intake 13-15 mg/Kg BW/day of placebo into 3 divided doses after meal as UDCA treatment group, till the endpoint or the 8th week.
  Arms: Placebo

SUMMARY:
Cholestatic drug-induced liver injury (DILI) is the severe form of DILI with a grave outcome. Drug-metabolizing enzymes play an important role in the metabolism of drugs. The genetic polymorphism of drug-metabolizing enzymes may influence the activities and expression of these enzymes and thereby affect the susceptibility and severity of DILI. UDP-glucuronosyltransferase (UGT) is an important phase 2 detoxification enzyme, which is related to congenital hyperbilirubinemia. Recently, the genetic polymorphism of UGT1A1 was reported to be associated with jaundice induced by some drugs, and UGT1A7 was shown to be related to the susceptibility of hepatocellular carcinoma and other cancers. Ursodeoxycholic acid (UDCA ) is a hydrophilic bile acid that is increasingly used for the treatment of various cholestatic disorders. The aims of this study are (1) to assess the association of the genetic polymorphism of UGT1A1 and 1A7, and the susceptibility and severity of drug-induced liver injury (DILI), with emphasis on the cholestatic DILI; (2) to evaluate the treatment effect of UDCA in the DILI, with special reference to the cholestatic hepatotoxicity.

DETAILED DESCRIPTION:
Cholestatic drug-induced liver injury (DILI) is the severe form of DILI with a grave outcome. Drug-metabolizing enzymes play an important role in the metabolism of drugs. The genetic polymorphism of drug-metabolizing enzymes may influence the activities and expression of these enzymes and thereby affect the susceptibility and severity of DILI. UDP-glucuronosyltransferase (UGT) is an important phase 2 detoxification enzyme, which is related to congenital hyperbilirubinemia. Recently, the genetic polymorphism of UGT1A1 was reported to be associated with jaundice induced by some drugs, and UGT1A7 was shown to be related to the susceptibility of hepatocellular carcinoma and other cancers. Ursodeoxycholic acid (UDCA ) is a hydrophilic bile acid that is increasingly used for the treatment of various cholestatic disorders. The aims of this study are (1) to assess the association of the genetic polymorphism of UGT1A1 and 1A7, and the susceptibility and severity of drug-induced liver injury (DILI), with emphasis on the cholestatic DILI; (2) to evaluate the treatment effect of UDCA in the DILI, with special reference to the cholestatic hepatotoxicity.

Owing to the limited number of DILI patients, 3 years are needed in this study. Each year, a total of 60 patients with DILI and 60 age- and sex-matched controls will be enrolled in this study. Their genetic polymorphisms of UGT1A1 and UGT1A7 will be assessed using the real time PCR, or PCR with RFLP. The DILI patients will be randomized to UDCA Treatment group and Control group. UDCA 13-15 mg/kg/day with 3 divided doses will be administered to the patients with Treatment group.

The frequencies of genotypes of UGT1A1 and 1A7 will be compared between DILI cases and controls, survival cases and non-survival cases, and cholestatic and non-cholestatic cases. Chi-square test, with or without Yates' correction, will be used to compare the categorical parameters. A paired t test will be performed to compare the continuous parameters. Odds ratios (OR) and confidence intervals (CI) will be calculated using a logistic regression analysis. The multivariate logistic regression analysis will be applied to check on the OR, adjusted with other possible risk factors. Survival rates will be estimated from survival curves based on the Kaplan-Meier method and compared with the log-rank test between the UDCA Treatment group and Control group.

We believe that this pharmacogenetic study may help us realize the pathogenesis of cholestatic DILI, and the clinical trial can elucidate the therapeutic value of UDCA in the DILI, especially in the cholestatic hepatotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Drug-induced liver injury, meet the DILIN criteria.

Exclusion Criteria:

* Other systemic diseases may cause elevation of liver enzymes: viral hepatitis, alcoholic liver disease, autoimmune hepatitis, primary biliary cirrhosis, Wilson's disease, hemochromatosis, congestive heart failure, hypoxia, sepsis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-04 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
severe degree drug-induced liver injury, fatality or liver transplantation | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Shin Huang, M.D., Principal Investigator — Taipei Veterans General Hospital, Taipei, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan